CLINICAL TRIAL: NCT06603779
Title: Integrated Neuromuscular Inhibition Versus Cervical and Scapular Stabilization Exercises on Myofascial Trigger Points of Upper Trapezius: Randomized Controlled Trial.
Brief Title: Integrated Neuromuscular Inhibition Versus Cervical and Scapular Stabilization Exercises on Myofascial Trigger Points of Upper Trapezius
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Dina Al-Amir Mohamed Hussein, Lecturer of Physical Therapy, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Beni-Suef University22
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Trigger Point Pain, Myofascial
MeSH Terms: conditions — Myofascial Pain Syndromes

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Integrated Neuromuscular Inhibition Group (Experimental): This group will receive the Integrated Neuromuscular Inhibition Technique which consists of ischemic compression, strain counter strain, and muscle energy technique
  Interventions: Other: Integrated Neuromuscular technique
- Cervical and Scapular Stabilization exercises Group (Experimental): This group will receive a group of exercises for the neck and scapula which will strengthen both of them
- Ultrasound Therapy Group (Placebo Comparator): This group will receive ultrasound Therapy
  Interventions: Device: Ultasound Therapy

INTERVENTIONS:
Device: Ultasound Therapy — a device that transmit ultrasound waves to the participant through direct contact
  Arms: Ultrasound Therapy Group
Other: Integrated Neuromuscular technique — Integrated Neuromuscular technique is a kind of Manual therapy which include Ischemic Compression, Strain counter-strain and muscle energy technique
  Arms: Integrated Neuromuscular Inhibition Group
Other: Cervical and Scapular Stabilization exercises — Cervical and Scapular Stabilization exercises are a group of therapeutic exercises.

SUMMARY:
This trial will involve three groups. The Integrated Neuromuscular Inhibition group will receive the integrated neuromuscular inhibition technique. The cervical and Scapular stabilization group will receive cervical and scapular stabilization exercises. The ultrasound group will receive ultrasound therapy

ELIGIBILITY:
Inclusion Criteria:

* Patients with active trigger points in the upper trapezius for more than 2 weeks based on the Simons Criteria.
* Age ranged from 18-25 years.
* Pain intensity ≥ 3 on VAS.
* Females and males.

Exclusion Criteria:

* Patients indicated for surgery.
* Patients with symptomatic disc lesions.
* Patients with rheumatological diseases or traumatic neck injury.
* Patients injected with corticosteroids in the last 6 months.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-07-28 (Actual); Study Completion 2025-07-28 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | 1-3 months
  Visual Analogue Scale is a scale that measures pain intensity. Subjects will instructed to indicate their current pain by marking a point on a 10 mm transverse line with 0 degrees meaning "no pain" and 10 meaning the "worst pain"
Pressure Pain Algometer | 1-3 months
  The pressure pain Algometer is a device that measures the pain threshold of the subjects.
Neck Pain and Disability Questionnaire (NDI) | 1-3 months
  Neck Pain and Disability is a questionnaire that measures neck pain and disabilities in subjects. Each question in the questionnaire will explained in detail and the subject will be asked to select one sentence out of six that best describes their function, a higher score indicates a great loss of function.
36-item Short-Form Health Questionnaire | 1-3 months
  36-item Short-Form Health Questionnaire will measure quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Banī Suwayf, Egypt